CLINICAL TRIAL: NCT06500988
Title: Patient Centered Mobile Health Technology-Enabled Atrial Fibrillation Management: Phase 2
Brief Title: Mobile Health Technology-Enabled AFib Management
Acronym: mTECH Afib
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Pharmaceutical Research & Manufacturers Of America Foundation (Unknown); Apple Inc. (Industry); Itamar-Medical, Israel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00453569
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation; Behavior
Keywords: Remote Patient Monitoring; Atrial Fibrillation; Risk Factor Modification; Digital Health; Mobile Health
MeSH Terms: conditions — Atrial Fibrillation; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corrie Virtual Atrial Fibrillation Management Program (Experimental): Multicomponent virtual atrial fibrillation management program
  Interventions: Combination Product: Corrie Virtual Atrial Fibrillation Management Program
- Usual Care (No Intervention): Receives usual care. Usual care is defined as care according to the patients care team's standard practice

INTERVENTIONS:
Combination Product: Corrie Virtual Atrial Fibrillation Management Program — Intervention aims to implement a comprehensive digital atrial fibrilation guideline-recommended toolkit
  Arms: Corrie Virtual Atrial Fibrillation Management Program

SUMMARY:
The overall objective of this proposal is to evaluate the effect on quality of life of a comprehensive digital atrial fibrillation (AFib) management tool that will empower patients to a) take an active role in learning about AFib management options, starting and adhering to evidence-based therapies and lifestyle changes and b) to guide the patients during AFib episodes which are associated with anxiety and impairment in quality of life.

Researchers plan to evaluate the effectiveness of this novel digital toolkit in improving quality of life and decreasing AFib burden in a randomized clinical trial (RCT). A pilot study assessing feasibility and retention of the intervention was previously conducted (NCT05400837)

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or older at time of consent
2. Diagnosis of paroxysmal (Afib lasting less than 7 days) or persistent (7 days or longer) atrial fibrillation
3. BMI (Body Mass Index) ≥ 27.0

Exclusion Criteria:

1. Permanent Afib (decision has been made not to attempt sinus rhythm)
2. Severe valvular disease
3. Moderate mitral valve stenosis
4. Prior cardiac surgery
5. Presence of implanted cardiac device
6. History of cardiac arrest
7. Left ventricular ejection fraction (LVEF) ≤ 35%
8. Life expectancy < 1 year
9. Non-English speaking
10. Treating clinician deems unsafe for exercise
11. Any other reason that makes patient unsuitable for study at the discretion of the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Quality of Life as measured by Atrial Fibrillation Effect on Quality-of-Life (AFEQT) survey | 6 months
  Measured by Atrial Fibrillation Effect on Quality-of-Life (AFEQT), which consists of 20 items. Score ranges from 0 to 100 with higher scores signifying better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: David Spragg, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Outpatient Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No